CLINICAL TRIAL: NCT06061471
Title: A Randomized, Double-blind, Phase II Clinical Study to Evaluate the Efficacy and Safety of AK111 in the Treatment of Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: To Evaluate the Efficacy and Safety of AK111 Injection in the Treatment of Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK111-203
Record Dates: First submitted 2023-09-24; First posted 2023-09-29 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Psoriasis; Skin Diseases
MeSH Terms: conditions — Psoriasis; Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: AK111 regimen 1 (Experimental)
  Interventions: Drug: AK111
- Experimental: AK111 regimen 2 (Experimental)
  Interventions: Drug: AK111

INTERVENTIONS:
Drug: AK111 — AK111 regimen 1-subcutaneous injection,until week 24.
  Arms: Experimental: AK111 regimen 1
Drug: AK111 — AK111 regimen 2-subcutaneous injection,until week 24.
  Arms: Experimental: AK111 regimen 2

SUMMARY:
This is a randomized, double-blind phase II clinical study to evaluate the efficacy and safety of AK111 in the treatment of subjects with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
This is a randomized, double-blind phase II clinical study to evaluate the efficacy and safety of AK111 in the treatment of subjects with moderate to severe plaque psoriasis. The study has 2 parts: first part (randomized double-blind) and second part (open).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥18 years old.
2. Subjects with moderate to severe plaque psoriasis with or without psoriatic arthritis.
3. At screening and baseline, PASI score ≥ 12, BSA ≥ 10%, sPGA ≥ 3.
4. Suitable for systematic therapy assessed by investigators.
5. Subjects who are women of childbearing potential must be practicing an adequate, medically acceptable method of birth control during the study and for at least 6 months after the last investigational drug administration.

Exclusion Criteria:

1. Types of psoriasis other than chronic plaque-type psoriasis.
2. Drug-induced psoriasis.
3. Evidence of active TB. Patients with evidence of latent tuberculosis may enter the trial after sufficient treatment had initiated and maintained according to protocol.
4. Positive results of confirmatory test for hepatitis B, hepatitis C, human immunodeficiency virus (HIV) or syphilis.
5. History of repeated chronic infection, had any serious infection or systemic infection within 2 months before screening.
6. Progressive or uncontrolled symptoms or signs of circulatory, respiratory, digestive, neuropsychiatric or psychological,hematological, endocrine and other systems before randomization.
7. History of malignant tumour within 5 years before screening.
8. Previous or current autoimmune diseases.
9. Allergic to any component of the investigational drug, or have had severe allergic reactions to monoclonal antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 454 (Actual)
Dates: Start 2023-09-22 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
The percentage of subjects who achieved at least 75% reduction in Psoriasis Area Severity Index （PASI）score from baseline (PASI 75) and the percentage of subjects with sPGA 0/1 at week 16. | at week 16
  PASI is a combined assessment of a lesion severity and affected area into a single score: 0 (no disease) to 72(maximal disease). The body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for a final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%),and severity is estimated by clinical signs, erythema, induration and desquamation: scale 0 (none) to 4 (maximum).Final PASI = sum of severity parameters for each area * area score weight of section (head: 0.1, arms: 0.2, body: 0.3,legs: 0.4).PASI 50, PASI75 and PASI 90 were defined as participants achieving >= 50%, >= 75% or >= 90% improvement from baseline, respectively.The sPGA is an instrument providing a subjective evaluation of the overall severity of psoriasis, based on severity of induration, scaling, and erythema. The scores are: 0 = clear; 1 = minimal; 2 = mild; 3 = moderate; 4 = marked; 5 =severe.

SECONDARY OUTCOMES:
The percentage of subjects who achieved at least 90% reduction in PASI score from baseline (PASI 90). | at week 16

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - The First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Affiliated Hospital of Chengde Medical University, Chengde, Hebei
  - Nanyang First People's hospital national third class a hospital, Nanyang, Henan
  - Yichang central People's hospital, Yichang, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The affiliated hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Dermatology hospital of Jiangxi province, Nanchang, Jiangxi
  - Tianjin academy of traditional Chinese medicine affiliated hospital, Tianjin, Tianjin Municipality
  - Hangzhou First People's hospital, Hangzhou, Zhejiang
  - The first hospital of Jiaxing, Jiaxing, Zhejiang

IPD SHARING:
Plan to Share IPD: No